CLINICAL TRIAL: NCT01918553
Title: Cohort Study on the Age-related Macular Degeneration: Incidence and Research for Predisposing Factors
Acronym: ECLAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2012/31
Record Dates: First submitted 2013-07-08; First posted 2013-08-07 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Elderly French Population; Age-related Macular Degeneration
Keywords: AMD; epidemiology; risk factors; cohort study
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subject in the study ALIENOR (Experimental)
  Interventions: Other: clinical parameters; Other: visual acuity exams; Other: retinophotography; Other: SD-OCT; Other: Intra ocular Pressure (IOP); Other: retinal imaging (OPTOMAP); Other: axial length (IOL master)

INTERVENTIONS:
Other: clinical parameters
Other: visual acuity exams
Other: retinophotography
Other: SD-OCT
Other: Intra ocular Pressure (IOP)
Other: retinal imaging (OPTOMAP)
Other: axial length (IOL master)

SUMMARY:
Age-related Macular Degeneration (AMD) is the most cause of blindness in the industrialised countries. There are few epidemiological studies on the incidence of this disease. Studying the incidence of AMD in an elderly French population and identifying the predisposing factors is very important to allow a major advance in the epidemiological knowledge of AMD. This study will contribute to the identification of the clinical, genetic and modifiable parameters associated at the risk of developing AMD. This could result in means prevention as well as in the identification of subjects as high risk of AMD

DETAILED DESCRIPTION:
Age-related Macular Degeneration is the most cause of blindness in the industrialised countries. There are few French epidemiological data on this disease. Worldwide, studies have included a small number of very old subjects. Thus, it is important to estimate the AMD incidence in an elderly French population, in order to evaluate more precisely the number of cases in the French population. Besides, some clinical, genetic and modifiable parameters predisposing to the AMD are under study. The aim of the ECLAIR project is to study the 8-year incidence of AMD in an elderly French population and to identify the predisposing factors. It is based on an existing cohort study (ALIENOR) in which some clinical, genetic and modifiable data were collected at baseline, 2 and 4 years. It is the only cohort study performed in France in this field since fifteen years in parallel with another one performed in Dijon according to the same methodology. It is important to extend the study to 8 years in order to have a sufficient statistical power for the identification of predisposing factors. In the ECLAIR study, there is no treatment. The subjects will be followed during 2 years (6 and 8 years after baseline of the Alienor study). The visit 1 (A0) will be the inclusion visit where the subjects will sign the inform consent and will perform ophthalmological examinations. The subjects will come back 2 years later for the visit 2 (A2). In this second visit, the ophthalmological examinations will be the same that is: measure of clinical parameters, measurement of visual acuity exams, retinophotography,spectral domain optical coherence tomography (SD-OCT), intraocular pressure, retinal imaging (OPTOMAP), axial length (IOL master)

ELIGIBILITY:
Inclusion Criteria:

* Subject participating in the study ALIENOR
* Affiliated to a social security
* Consent signed by the patient and the investigator

Exclusion Criteria:

- Health incompatible with one hour and a half ophthalmic examination

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
8-year incidence of late AMD (neovascular and/or atrophic) | at day 0 (inclusion in ECLAIR study and 6 years after inclusion in ALIENOR cohort) and year 2 after inclusion (end of ECLAIR study and 8 years after inclusion in ALIENOR cohort)

SECONDARY OUTCOMES:
best-corrected visual acuity (ETDRS methodology) measured in visit 1 and 2 years later with ETDRS methodology | at day 0 (inclusion) and year 2 after inclusion (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Korobelnik Jean-François, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Unité Médicale Rétine Neuro-Ophtalmologie - Service d'Ophtalmologie - Hopital Pellegrin, Bordeaux, France

REFERENCES:
- [Background] Cougnard-Gregoire A, Delyfer MN, Korobelnik JF, Rougier MB, Malet F, Le Goff M, Dartigues JF, Colin J, Barberger-Gateau P, Delcourt C. Long-term blood pressure and age-related macular degeneration: the ALIENOR study. Invest Ophthalmol Vis Sci. 2013 Mar 28;54(3):1905-12. doi: 10.1167/iovs.12-10192. PMID 23404120
- [Background] Merle B, Delyfer MN, Korobelnik JF, Rougier MB, Colin J, Malet F, Feart C, Le Goff M, Dartigues JF, Barberger-Gateau P, Delcourt C. Dietary omega-3 fatty acids and the risk for age-related maculopathy: the Alienor Study. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):6004-11. doi: 10.1167/iovs.11-7254. PMID 21705687
- [Background] Delcourt C, Delyfer MN, Rougier MB, Amouyel P, Colin J, Le Goff M, Malet F, Dartigues JF, Lambert JC, Korobelnik JF. Associations of complement factor H and smoking with early age-related macular degeneration: the ALIENOR study. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5955-62. doi: 10.1167/iovs.10-6235. PMID 21642625